# Title: The Efficacy of Adjuvant Oral Care in Prevention of Ventilator-Associated Pneumonia

- ClinicalTrials.gov Identifier
  - o NCT06039995
- Study Design
  - Randomized Controlled Trial
- Sponsor / Responsible Party
  - o University of Health Sciences
- Study Site
  - o Services Hospital, Lahore, Pakistan
- Principal Investigator
  - Akash Samuel
    - University of Health Sciences
- Document Type
  - Statistical Analysis Plan (SAP)
- SAP Version
  - o Version 1.0
- Document Date
  - o 15 December 2025

### **Statistical Analysis Plan (SAP)**

#### Analysis Population

 All randomized participants (n=100) were included in the analysis, with 50 patients in each study arm. No attrition was reported.

### Descriptive Statistics

- Continuous variables (age, ICU stay) were summarized using means and standard deviations.
- Categorical variables (sex, VAP incidence, mortality) were summarized using frequencies and percentages.

#### Primary Outcome Analysis

 $_{\odot}$  The incidence of VAP was compared between intervention and control groups using a chi-square test or Fisher's exact test, as appropriate. The level of statistical significance was set at p < 0.05.

### Secondary Outcome Analyses

- Duration of ICU Stay: Compared between groups using an independent-samples
  t-test, assuming approximate normality.
- Mortality Rates: Compared using chi-square analysis.

# Assumptions and Verification

- Normality assumptions for continuous outcomes were assessed using descriptive distribution checks.
- o Equality of variances was evaluated prior to parametric testing.
- No adjustments for multiple comparisons were applied, as secondary outcomes were exploratory.

# • Handling of Missing Data

 No missing outcome data were reported; therefore, no imputation methods were required.

# Safety Analysis

 Adverse events were summarized descriptively. Serious and non-serious adverse events were compared between groups. No intervention-related adverse events were reported.